CLINICAL TRIAL: NCT04867551
Title: A Phase II Clinical Study of KDT-3594 in Japanese Patients With Early Parkinson's Disease
Brief Title: A Clinical Study of KDT-3594 in Japanese Patients With Early Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDT1202A
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KDT-3594 (Experimental)
  Interventions: Drug: KDT-3594

INTERVENTIONS:
Drug: KDT-3594 — oral administration, dose titration

SUMMARY:
Objective of this study is to investigate the safety, pharmacokinetics and efficacy of KDT-3594 in patients with early Parkinson's disease without a concomitant medication of L-dopa.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients
* Patients who are diagnosed with Parkinson's disease according to UK Parkinson's Disease society brain bank clinical diagnostic criteria
* Patients with Parkinson's disease in Stages 1 to 3 on the Modified Hoehn and Yahr Scale

Exclusion Criteria:

* Patients who are suspected any parkinsonism except for idiopathic Parkinson's disease.
* Patients who underwent neurosurgical treatment (stereotaxic destruction, deep brain stimulation etc.) for PD, or patients for whom surgical treatment is scheduled during the study
* Patients with a complication of obvious dementia, or patients with Mini-Mental State Examination (MMSE) score < 24 points

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | 8 weeks
  The numbers of events and subjects, the incidence regarding adverse events.
Plasma concentrations of KDT-3594 and its metabolites | 8 weeks
  Plasma concentrations of KDT-3594 and its metabolites during treatment period.

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 8 weeks
  Change from baseline (Week 0) in MDS-UPDRS total score

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No